CLINICAL TRIAL: NCT00754780
Title: Phase II Clinical Trial of Pirfenidone for the Treatment of Patients With Neurofibromatosis Type I
Brief Title: Clinical Trial of Pirfenidone in Adult Patients With Neurofibromatosis 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Dusica Babovic-Vuksanovic, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1835-99; MC0077; Mayo Pirfenidone Study
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Neurofibromatosis
Keywords: NF1; plexiform neurofibroma
MeSH Terms: conditions — Neurofibromatoses; Neurofibroma, Plexiform | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pirfenidone — Capsule 800 mg TID, oral

SUMMARY:
The study is a phase II, open label trial of oral Pirfenidone in 24 adult patients with neurofibromatosis type 1.

Pirfenidone is a new, broad-spectrum anti-fibrotic drug, with proven in vitro and in vivo negative effects on fibroblast growth and collagen matrix synthesis. Human studies indicate promising therapeutic effects in arresting and reversing fibrosis in a variety of different conditions, where the excessive formation of fibrous tissue is a major pathogenic mechanism. Since the fibrous tissue is a significant component of neurofibroma, reduction of fibrosis could diminish tumor progression and lead to tumor shrinkage. Therefore, Pirfenidone is an excellent candidate for the treatment of plexiform neurofibromas and surgically unresectable tumors in patients with NF1.

DETAILED DESCRIPTION:
Specific aims of this study are:

1. To evaluate efficacy of Pirfenidone in NF1 patients with disfiguring or disabling plexiform neurofibroma (PN) and spinal neurofibromas (SN)
2. To determine the acute, subacute and chronic toxicity of Pirfenidone in patients with NF1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neurofibromatosis type I, based on clinical criteria (NIH Consensus Development Conference, 1988). Tumors will not be confirmed histologically, since the biopsy could cause a change in tumor growth and such interfere with effect of Pirfenidone treatment.
* Male or female patients
* Age 18 years old
* All patients should be mentally capable of signing the consent form or should have a legal guardian to provide consent
* Patients who are experiencing symptoms from neurofibromatous lesions and who refuse surgery or are not good surgical candidates, such as those with plexiform neurofibroma who are experiencing significant discomfort, disfigurement or nerve compression or
* Presence of multiple spinal neurofibromas in which the surgical removal would carry a major risk for spinal cord damage.

Exclusion Criteria:

* Tumors for which surgical removal could lead to permanent (or long-term) relief of symptoms
* Patients with open skin lesions and patients for whom surgery is being contemplated or who had surgery less than 4 weeks from starting treatment
* Patients for whom biopsy is warranted for suspected malignancies
* Individuals younger than 18 years
* Pregnant and lactating women
* Inability to have MR imaging (e.g. claustrophobia, pacemaker or allergy to contrast dye, if administration is needed for neurofibroma imaging)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2000-09; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
tumor volume | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dusica Babovic-Vuksanovic, M.D., Principal Investigator — Mayo Clinic